CLINICAL TRIAL: NCT01691170
Title: Quadriceps Femoris Strengthening Versus Hamstring Stretching for Patellofemoral Pain Syndrome: A Randomized Clinical Trial.
Brief Title: Comparison of Two Protocols for Patellofemoral Pain Syndrome
Acronym: PFPS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Gabriel Peixoto Leão Almeida, PT, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USP01
Record Dates: First submitted 2012-09-16; First posted 2012-09-24 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Pattelofemoral pain syndrome; Stretching; Strengthening
MeSH Terms: conditions — Patellofemoral Pain Syndrome

ARMS (2):
- Quadriceps Strengthening (Active Comparator)
  Interventions: Other: Quadriceps Strengthening
- Stretching Hamstring (Active Comparator)
  Interventions: Other: Stretching Hamstring

INTERVENTIONS:
Other: Stretching Hamstring
  Arms: Stretching Hamstring
Other: Quadriceps Strengthening
  Arms: Quadriceps Strengthening

SUMMARY:
The patellofemoral pain syndrome (PFPS) is defined as a painful complaint in the anterior aspect of the knee, although peripatellar pain and / or retropatellar are also common. In general, conservative treatment is the initial option of choice for patients with PFPS, however, the lack of a specific causal factor makes it difficult to choose the best treatment so early. This way, the purpose of this study is investigate the effects of the quadriceps femoris strengthening versus hamstring stretching in patients with pattellofemoral pain.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of anterior knee pain for at least 1 moth;
* Average pain level of 3 or more on a 10-cm visual analogue scale during stepping up and down a 25-cm height;
* Anterior or retropatellar knee pain on at least 2 of the following activities: prolonged sitting, climbing stairs, squatting, running, kneeling, and hopping/jumping;
* Presence of 2 of the following clinical criteria on assessment: pain during apprehension test, pain during the patellar compression test, and crepitation during the compression test.

Exclusion Criteria:

* Previous knee surgery or arthritis;
* History of patellar dislocation or subluxation, malalignment, or ligament laxity;
* Patellar tendon pathology or chondral damage;
* Spinal referred pain;
* History of other abnormalities such as leg length inequalities (>2 cm);
* Medication as a part of the treatment;
* Previous physical therapy or acupuncture treatment for the knee within the previous 30 days.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2011-02 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Participants will be followed for the duration of 8 weeks.
  Pain was assessed using an 11-point numeric pain rating scale (NPRS), on which 0 denoted an absence of pain and 10 denoted unbearable pain.

SECONDARY OUTCOMES:
Lysholm Scale | Participants will be followed for the duration of 8 weeks.
  This questionnaire is made up of eight items with objective response options. The final score is expressed in nominal and ordinal form, as follows: 95 to 100 points - excellent; 84 to 94 points - good; 65 to 83 points - fair; and 64 or fewer points - poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Speech and Occupational Therapy Department, University of São Paulo., São Paulo, São Paulo, Brazil